CLINICAL TRIAL: NCT06947850
Title: TITLE: Toyos Clinic / A Phase 4 Study to Assess Longer Duration of Treatment With Cenegermin in Moderate to Severe Dry Eye-Associated Neurotrophic Keratitis
Brief Title: DOMPE -MT Neurotrophic Keratitis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Toyos Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMT-2021-02
Record Dates: First submitted 2025-04-17; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Dry Eye; Neurotrophic Keratitis
Keywords: dry eye; Neurotrophic Keratitis
MeSH Terms: conditions — Dry Eye Syndromes | interventions — cenegermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 8 week cenegermin treatment (Active Comparator): All participants receive cenegermin topical ophthalmic drops 20mcg/ml six times daily for a treatment period of either 8 or 16 weeks followed by a follow up period total52 weeks total for each study arm.
  Interventions: Drug: Cenegermin Ophthalmic Solution [Oxervate]
- 16 week cenegermin (Active Comparator): All participants receive cenegermin topical ophthalmic drops 20mcg/ml six times daily for a treatment period of either 8 or 16 weeks followed by a follow up period total52 weeks total for each study arm.
  Interventions: Drug: Cenegermin Ophthalmic Solution [Oxervate]

INTERVENTIONS:
Drug: Cenegermin Ophthalmic Solution [Oxervate] — Oxervate (cenegermin-bkbj) is commonly used to treat neurotrophic keratitis

SUMMARY:
TITLE: Toyos Clinic / A Phase 4 Study to Assess Longer Duration of Treatment with Cenegermin in Moderate to Severe Dry Eye-Associated Neurotrophic Keratitis

ELIGIBILITY:
Inclusion Criteria:1. Provision of signed and dated informed consent form and HIPPA authorization.

2. Stated willingness to comply with all study procedures and availability for the duration of the study 3. Male or female, aged 18 to 85. 4. Subjects with moderate to severe ocular pain defined as SANDE questionnaire score of >25 mm at time of screening not due to causes other than dry eye associated with NK in the opinion of the investigator.

5. Have used and/or desired to use an artificial tear substitute for dry eye symptoms in the past 3 months.

6. Have normal lid anatomy. 7. For females of reproductive potential:use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.

8. For males of reproductive potential:use of condoms or other methods to ensure effective contraception with partner 9. Are postmenopausal (no menstrual cycle for at least one year prior to Visit 1) or have undergone bilateral tubal ligation, hysterectomy, hysterectomy with uni- or bilateral oophorectomy, or bilateral oophorectomy.

10. Patients with stage 1 NK characterized by epithelial irregularity most commonly in the form of punctate keratopathy without epithelial defect or Stage 2 (persistent epithelial defect, PED).

11. PED or corneal ulceration of at least 2 weeks duration refractory to one or more conventional non-surgical treatments for neurotrophic keratitis (e.g., preservative-free artificial tears, gels or ointments; discontinuation of preserved topical drops and medications that can decrease corneal sensitivity; therapeutic contact lenses).

12. Evidence of decreased corneal sensitivity (≤ 4 cm using the Cochet-Bonnet aesthesiometer) within the area of the PED or corneal ulcer and outside of the area of the defect in at least one corneal quadrant.

13. BCDVA of 20/200 or better by Snellen or >/=0.1 decimal units.

-

Exclusion Criteria:

1. Have a known hypersensitivity or contraindication to the investigational product or their components.
2. Severe systemic allergy.
3. Topical glaucoma medications or oral medications that are not being taken at a stable dose for the past 90 days.
4. Topical dry eye medications within the last month except unpreserved artificial tears which will be allowed throughout the study as needed.
5. Active viral, fungal or bacterial infection or active intraocular inflammation.
6. Subjects must be unwilling to abstain from eyelash growth medications for the duration of the trial.
7. Subjects must not have had penetrating intraocular surgery, refractive surgery or corneal transplantation, eyelid surgery within 12 weeks prior to Visit 1.
8. Febrile illness within one week of screening visit.
9. Treatment with another investigational drug or other investigational intervention withinone month of screening visit.
10. Have serious or severe disease or uncontrolled medical condition that in the judgment of the investigator could confound study assessments or limit compliance.
11. Subjects that are currently pregnant or intend to become pregnant during the course of the study, are breastfeeding, or who are unwilling to use highly effective birth control measures such as hormonal contraceptives, and/or mechanical barrier methods during the course of the trial.
12. Use of contact lenses during trial.
13. Amniotic membranes within two weeks prior to screening.
14. Punctal plugs will be allowed as long as they have remained stable for at least 90 days.
15. No neurostimulation including varencicline, acupuncture or TrueTear or like devices within one month of screening.

    -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-21 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
TITLE: Toyos Clinic / A Phase 4 Study to Assess Longer Duration of Treatment with Cenegermin in Moderate to Severe Dry Eye-Associated Neurotrophic Keratitis | 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Toyos Clinic, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided